CLINICAL TRIAL: NCT05128812
Title: Study of the Anxiolytic Effects, Improvement of Sleep Quality and Bioparametric Measures in Individuals Taking an Extract of Lippia Citriodora.
Brief Title: Study of the Effects of Plx on Bioparametric Measurements.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Assistant Professor, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UA-2021-03-26
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Quality of Life; Antidepressive Agents; Depression, Anxiety; Sleep Initiation and Maintenance Disorders; Body Composition; Stress, Psychological
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (Placebo Comparator): Nutraceutical placebo intake group
  Interventions: Dietary Supplement: PLX
- PLX400mg GROUP (Experimental): Intake of natural herbal dietary supplement composed of lemon verbena extract (Lippia citriodora).
  Interventions: Dietary Supplement: PLX

INTERVENTIONS:
Dietary Supplement: PLX — Intake of natural food supplement of vegetable origin based on lemon verbena extract (Lippia citriodora). To study the anxiolytic effects in subjects with high perceived stress levels and low sleep quality.

SUMMARY:
The main objective is to study the effects of the intake of a nutraceutical on health indicators, focused on sleep and stress, as well as cardiovascular (blood pressure...), circulating (cortisol) and body composition parameters in a Spanish adult population.

DETAILED DESCRIPTION:
Anxiety is a normal part of life, and generally is a temporary condition. However, anxiety can occasionally prolong in time, having an impact on everyday activities, and give rise to other conditions, such as depression, drug abuse, cardiovascular disease, and insomnia. There are a number of synthetic drugs that are commonly used to treat anxiety. These are mainly antidepressants and benzodiazepines. However, their high cost, important side effects and a rising interest in natural solutions have driven researchers to search for botanical-based formulas. To this end, there are a number of plants that have been described to possess potential sedative and anxiolytic effects. Of note is lemon verbena (Lippia citriodora), which is native of Western South America but is also cultivated in the Mediterranean region and Middle East.

ELIGIBILITY:
Inclusion Criteria:

1. Over 21 years of age;
2. Without any chronic pathology;
3. Score on the Spielberg Trait-State Anxiety Inventory (STAI-S) comprising 20 items, greater than 40 (probable clinical levels of anxiety);
4. Pittsburgh Sleep Quality Index (PSQI) score greater than 5 (poor sleep quality).

Exclusion Criteria:

* Failure to meet the inclusion criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
WEIGHT | 3 months
  The weight of the subjects will be obtained using the TANITA (Tokyo, Japan).
HEIGHT | 3 months
  The height of the subjects will be measured with the SECA 123 stadiometer (Hamburg, Germany).
BLOOD PREASURE | 3 months
  Measurement of blood pressure (systolic and diastolic) with a digital tensiometer.
FAT MASS | 3 months
  Assessment of body composition using the TANITA (Tokyo, Japan) validated bioimpedance scale to obtain the results of fat mass.
VISCERAL FAT | 3 months
  Assessment of body composition using the TANITA (Tokyo, Japan) validated bioimpedance scale to obtain the results of visceral fat.
BLOOD CORTISOL | 3 months
  Cortisol levels in blood by blood analysis.
SLEEP QUALITY | 3 months
  Measurement of sleep quality using the Pittsburgh sleep quality index.
STRESS | 3 months
  Measurement of perceived stress using the Perceived Stress Scale (PSS).
ANXIETY | 3 months
  Measurement of perceived anxiety using the Spielberger Trait-State Anxiety Inventory questionnaire; it is an instrument created with the objective of assessing anxiety in two dimensions, state and trait.
PERCEIVED QUALITY OF LIFE | 3 months
  Measurement of quality of life using the World Health Organization Quality of Life (WHOQOL-BREF). The WHOQOL-BREF instrument provides a profile of quality of life, with each dimension or domain being scored independently. each dimension or domain scored independently. The higher the higher the score in each domain, the better the quality of life profile of the person being the person being assessed.
HEART RATE | 3 months
  An electrocardiogram is used to obtain the heart rate.
SLEEP HOURS | 3 months
  Use of a FITBIT device to monitor the hours of sleep of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Martinez Rodriguez, Assistant, Principal Investigator — Alicante University
Locations (1):
- University of Alicante, Alicante, Spain